CLINICAL TRIAL: NCT05578989
Title: The Effect of Virtual Reality Glasses Applied During Episiotomy on Pain and Satisfaction: Single Blind Randomized Controlled Trial
Brief Title: The Effect of Virtual Reality Glasses Applied During Vaginal Incision Suturing on Pain and Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Merva Orhan, MSc Midwife, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 135790
Record Dates: First submitted 2022-07-19; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Episiotomy; Dehiscence
Keywords: Obstetrics; Episiotomy; Virtual reality; Pain; Satisfaction
MeSH Terms: conditions — Pain; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group watching video with virtual reality glasses (Experimental): Women in the intervention group watched a video with virtual reality glasses during the episiotomy. (25 women)
  Interventions: Device: Virtual reality glasses
- Comparisongroup that does not use virtual glasses (No Intervention): The women in the control group were treated with without watching videos during the episiotomy. (25 women)

INTERVENTIONS:
Device: Virtual reality glasses — watching a video with music with virtual reality glasses.
  Arms: Group watching video with virtual reality glasses

SUMMARY:
The research was conducted as a randomized controlled clinical study to determine the effect of virtual reality glasses on pain and patient satisfaction during the episiotomy repair procedure. The sample consisted of 50 pregnant woman of whom 25 were in the control group and 25 were determined by randomization among primiparous pregnant woman who met the reasearch's criteria and agreed to participate in the study.

DETAILED DESCRIPTION:
Objective: The research was conducted as a randomized controlled clinical study to determine the effect of virtual reality glasses on pain and patient satisfaction during the episiotomy repair procedure.

Method: The research population consisted of 50 primiparous pregnant women who applied to the delivery room of Necip Fazıl City Hospital Gynecology and Child Additional Service Building between 15 June 2021 and 15 December 2021 for vaginal delivery. Data were collected with the Mother Identification Form and Visual Analogum Scales (VAS) Pain - Satisfaction Evaluation Forms. During the episiotomy repair procedure, 5 ml of lidocaine was administered to the patients in the intervention group; A video with music was watched with virtual reality glasses for an average of 10 minutes, just before starting the process and throughout the process. No application was made to the mothers in the control group, except for 5 ml of lidocaine, which was applied during episiotomy repair. In the evaluation of the data, mean, standard deviation, percentage and number values are given. Student's t test was used to compare normally distributed variables in two groups, and Mann Whitney U test was used to compare non-normally distributed variables in two groups. In testing the variables in different groups and times, repeated measures of variance analysis were applied. Relationships between categorical variables were tested with CI-square test, and relations between non-normally distributed numerical variables were tested with Spearman rank correlation coefficient. SPSS 22.0 Windows version package program was used in the analysis. P<0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 18-49
* Speak and understand Turkish
* Volunteering to participate in the study
* Being a primiparous (first-time woman) pregnant
* Being in the low pregnancy risk group without obstetric complications (bleeding, unreliable fetal heart rate…) at all stages of delivery
* To have given spontaneous delivery with a medio-lateral episiotomy incision in the hospital at the time of the study.
* Not having vision, hearing and perception problems
* No diagnosis or history of mental illness
* Not having any signs of infection such as vaginal redness, swelling
* Not be allergic to latex and local anesthetic drugs
* No communication problem,

Exclusion Criteria:

* Apgar score <7 in 1 minute and 5 minutes
* Having a neonatal anomaly
* Unusual use of lidocaine during episiotomy repair (lidocaine greater than 5 ml 2%)
* Those who did not meet the inclusion criteria, did not fill out the form and stopped participating in the study.
* Those with headaches

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-08-02 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | 10-15 munites.
  It is a scale used to measure subjective experiences. In the form of a 0-10 cm ruler, one end of the scale indicates 0 painlessness and the other end 10 indicates the most severe degree of pain intensity. The degree of pain intensity was evaluated by marking the pain perceived by the woman on the ruler.

SECONDARY OUTCOMES:
Visual Analogue Scale | 5 munites.
  It is a scale used to measure subjective experiences. It was used to assess satisfaction after episiotomy. One end of the scale, in the form of a 0-10 cm ruler, indicates dissatisfaction at all, and the other end of 10 indicates the highest degree of satisfaction. The satisfaction level of the woman was evaluated by marking the number on the ruler. Satisfaction was measured in the first 1-hour period immediately after the episiotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Aysel Bülez, Assist. Prof., Study Chair — Kahramanmaraş Sütçü İmam University institute of health sciences.
Locations (1):
- Necip Fazıl City Hospital/ Gynecology and Children, Kahramanmaraş, Turkey (Türkiye)